CLINICAL TRIAL: NCT02765256
Title: Fundamental Modification of the Gut Microbiota in the Treatment of Refractory Crohn's Disease
Acronym: Holiday
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Lindsey Albenberg, Assistant Professor of Pediatrics, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 823635
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Fluconazole; Vancomycin; Neomycin; Ciprofloxacin; polyethylene glycol 3350; Promethazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluconazole (Experimental): Vancomycin 500 mg oral suspension four times daily (Day 1-14), plus neomycin 1000 mg orally three times daily (Days 1-3), plus ciprofloxacin 750 mg orally twice daily (Day 4-14), plus Polyethylene Glycol 3350 (Miralax) 238 g dissolved in 64 ounces of Gatorade or Crystal Lite on day 2, plus fluconazole 400 mg orally once daily (Day 1-14). PRN (as needed) Promethazine 12.5mg up to every four hours (Days 1-3).
  Interventions: Drug: Fluconazole; Drug: Vancomycin; Drug: Neomycin; Drug: Ciprofloxacin; Drug: Polyethylene Glycol 3350; Drug: Promethazine
- Placebo (Placebo Comparator): Vancomycin 500 mg oral suspension four times daily (Day 1-14), plus neomycin 1000 mg orally three times daily (Days 1-3), plus ciprofloxacin 750 mg orally twice daily (Day 4-14), plus Polyethylene Glycol 3350 (Miralax) 238 g dissolved in 64 ounces of Gatorade or Crystal Lite on day 2, plus placebo for fluconazole. PRN (as needed) Promethazine 12.5mg up to every four hours (Days 1-3).
  Interventions: Drug: Vancomycin; Drug: Neomycin; Drug: Ciprofloxacin; Drug: Polyethylene Glycol 3350; Drug: Promethazine; Drug: Fluconazole placebo

INTERVENTIONS:
Drug: Fluconazole — 400mg orally once daily (Day 1-14)
  Other Names: Diflucan
  Arms: Fluconazole
Drug: Vancomycin — 500mg oral suspension 4 times daily (Day 1-14)
  Other Names: Vancocin
Drug: Neomycin — neomycin 1000 mg orally three times daily (Days 1-3)
  Other Names: Neo-Fradin
Drug: Ciprofloxacin — ciprofloxacin 750 mg orally twice daily (Day 4-14)
  Other Names: Cipro
Drug: Polyethylene Glycol 3350 — 238 g dissolved in 64 ounces of Gatorade or Crystal Lite on day 2
  Other Names: Miralax
Drug: Promethazine — PRN (as needed) Promethazine 12.5mg up to every four hours (Days 1-3).
  Other Names: Phenergan
Drug: Fluconazole placebo — Once daily
  Arms: Placebo

SUMMARY:
To determine the effect of a novel gut microbiota-targeted therapeutic regimen (bowel lavage and antibiotics with or without an antifungal) in the management of active Crohn's Disease (CD) that is refractory to conventional, immunosuppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant is capable of giving informed consent
* Males or females 18-75 years of age
* Normal kidney function (defined by normal serum creatinine [male: <1.27 mg/dL; female: <1.03 mg/dL])
* Normal aspartate aminotransferase [AST] (<41 U/L), alanine aminotransferase [ALT] (<63 U/L), and alkaline phosphatase (<126 U/L)
* Active CD defined as HBI ≥ 7
* CRP > 5 mg/dL or hs-CRP > 10mg/L (or 1mg/dL) or fecal calprotectin (FCP) > - - 350 mcg/g (within one month of enrollment)
* Have been treated with one of the following therapies** for at least 8 weeks with primary nonresponse or an initial response, followed by loss of response [LOR] (self-reported worsening of symptoms for ≥ 7 days): azathioprine, 6-mercaptopurine, methotrexate, adalimumab, certolizumab, golimumab, infliximab, natalizumab, vedolizumab, or ustekinumab **These medications must have been administered at standard, therapeutic dosages.

Exclusion Criteria:

* Known or suspected stricturing disease producing obstructive symptoms
* Active Clostridium difficile infection
* Unwillingness to provide informed consent
* Allergy or intolerance to the medications used in this study
* History of kidney disease
* History of liver disease
* Pregnant or lactating females
* Baseline QTc interval on EKG > 430 in males or > 450 in females
* Participants who, in the opinion of the investigator, may be non-compliant with study schedules or procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Albenberg, DO, Principal Investigator — University of Pennsylvania; James D Lewis, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluconazole | Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluconazole | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Median (Full Range); unit: years] | 44 [26 to 54] | 32.5 [20 to 66] | 39.5 [20 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 4 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Disease Activity by Harvey Bradshaw Index
Description: The primary endpoint will be the change in disease activity, as measured by Harvey-Bradshaw Index (HBI) score, between the enrollment visit and Day 15. All participants who withdraw for any reason prior to day 15 will be considered treatment failures. The HBI is a clinical score where points are given for each category below plus number of liquid bowel movements in previous day. A score of 3 or lower is considered remission. A score of 8 or higher is considered severe disease.
  General Well Being Very well 0 points Slightly below par 1 point Poor 2 points Very poor 3 points Terrible 4 points
  Abdominal Pain None 0 points Mild 1 point Moderate 2 points Severe 3 points
  Abdominal Mass None 0 points Dubious 1 point Definite 2 points Definite and tender 3 points
  Complications None 0 points Arthralgias +1 point Uveitis +1 point Erythema Nodosum + 1 point Aphthous ulcers +1 point Pyoderma Gangrenosum + 1 point Anal fissure + 1 point New fistula + 1
Time Frame: enrollment visit (baseline) and 15 days
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 4
score on a scale | -5 [-7 to 0] | -3 [-8 to -2]

2. Primary Outcome: Change in Disease Activity by Fecal Calprotectin (FCP)
Description: The second primary outcome measure will be the change in disease activity, as measured by fecal calprotectin, between the enrollment visit and day 15. The fecal calprotectin is a stool test which measures intestinal inflammation.
Time Frame: enrollment visit (baseline) and 15 days
Measure: Median (Full Range); unit: mcg/g
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 4
mcg/g | -16.5 [-116.48 to 94] | -380.5 [-1234 to -1]

3. Secondary Outcome: The Change in High-sensitivity C-reactive Protein (hsCRP)
Description: A secondary outcome measure will be the change in high-sensitivity C-reactive protein between the enrollment visit and day 15. The high-sensitivity C-reactive protein is a blood test which measures systemic inflammation.
Time Frame: enrollment visit (baseline) and 15 days
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 4
mg/dL | 4.1 [1.1 to 8.3] | -2 [-2.9 to 1.6]

4. Secondary Outcome: Safety and Tolerability of the Treatment Regimen Based on Medication Side Effects and/or Adverse Events (AEs).
Description: Number of Medication Side Effects and/or Adverse Events (AEs)
Time Frame: 105 days
Measure: Number; unit: Events
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 4
Events | 31 | 12

ADVERSE EVENTS:
Time Frame: 105 days
Arm/Group | Fluconazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluconazole (N=4) | Placebo (N=4)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Increased diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perianal irritation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decreased appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Defecation urgency (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruitment was difficult due to intensive methods with large number of/frequent study visits required. Small sample size is a major limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT02765256/Prot_SAP_000.pdf